CLINICAL TRIAL: NCT01709032
Title: Pilot Study of Deferasirox and Deferiprone Combination Oral Chelation for Individuals With Transfusion Dependent Thalassemia and High Iron Burden
Brief Title: Combination Deferasirox and Deferiprone for Severe Iron Overload in Thalassemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: The Cooley's Anemia Foundation, (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-009449
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-02

CONDITIONS: Thalassemia Major With Severe Transfusional Iron Overload
Keywords: Thalassemia; Chelation; Transfusion; Safety
MeSH Terms: conditions — Thalassemia | interventions — Deferasirox; Deferiprone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deferasirox and deferiprone (Experimental)
  Interventions: Drug: Deferasirox and deferiprone

INTERVENTIONS:
Drug: Deferasirox and deferiprone
  Other Names: Exjade; Ferriprox

SUMMARY:
We hypothesize that the combination treatment with deferasirox and deferiprone will be well tolerated and will result in significant improvement in cardiac and liver iron levels.

DETAILED DESCRIPTION:
Death and disability from iron related damage to the heart remain the most serious issue facing transfusion-dependent patients with thalassemia. However, over the past decade there have been several reports of improved survival and fewer cardiac complications. This improvement may be related to the availability of three chelators and also the accurate measurement of iron stores in various organs (e.g. heart and liver) with magnetic resonance imaging, which allows for personalized, tailored medical care for patients. The chelator characteristics, side effect profiles, and ability to remove iron from specific organs differ among the chelators, suggesting that combination therapy may be beneficial. Using two drugs at lower doses may be more tolerable than escalating doses of a single drug and may improve iron removal. The combination of deferoxamine and deferiprone has been shown to be particularly beneficial for reducing cardiac iron, but it requires a painful injection/infusion, which hinders adherence. This pilot study aims to investigate the safety of an oral-only combination chelator regimen (deferasirox and deferiprone) in individuals with thalassemia major with poorly controlled iron overload and to assess how well this chelator combination lowers iron stores over one year.

ELIGIBILITY:
Inclusion Criteria:

* Alpha or beta thalassemia
* Receiving chronic transfusions (at least 20 transfusions in lifetime) with iron overload requiring treatment with chelation
* Serum ferritin >500 ng/ml
* Liver iron concentration equal to or greater than 10 mg/g dw (by R2 MRI) or 7 to 10 mg/g dw (by R2 MRI) and not improving OR cardiac T2* between 6 and <20 ms
* Women of childbearing age must have a negative pregnancy test
* Agree to use approved method of contraception for the duration of the study
* Subjects must have a good understanding of the study and be willing to comply with study procedures

Exclusion Criteria:

* Subjects with past history of unexplained neutropenia (ANC < 1500/mcL), clinically significant renal disease (creatinine above the upper limit of normal), proteinuria >300 mg/L, clinically significant liver disease (ALT > 5x upper limit of normal), pulmonary or cardiovascular disease
* History of other clinically relevant oral, endocrine, neurologic, psychiatric, immunologic, bone marrow or skin disorder that contraindicates dosing with deferasirox or deferiprone
* History of adverse reaction or known allergy to either deferasirox or deferiprone necessitating drug discontinuation
* Currently receiving treatment for active hepatitis
* Use of any investigational agent in the past 30 days
* Cardiac T2* <6 ms, left ventricular ejection fraction < 56%, and/or arrhythmia (certain subjects may be eligible if they have already had a trial of deferoxamine and deferiprone). Subjects who refuse to use deferoxamine after extensive consultation with at least 2 health care providers will also be allowed to participate.
* Pregnant or breastfeeding females
* Unwilling or unable to comply with study related procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2017-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet L Kwiatkowski, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- Deferasirox and Deferiprone: Deferasirox and deferiprone
Period: Overall Study
Arm/Group | Deferasirox and Deferiprone
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Deferasirox and Deferiprone
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Liver Iron Concentration
Description: Determine the safety of the combination of Deferasirox and Deferiprone for the treatment of subjects with Thalassemia Major and Severe Iron Overload by assessing change in liver iron concentration from baseline to follow-up
Time Frame: 12 months
Population: Number with participants with improvement in liver iron concentration
Measure: Count of Participants; unit: Participants
Arm/Group | Deferasirox and Deferiprone
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: Number of Participants With Improvement in Cardiac T2* MRI
Description: Improvement in Cardiac T2* MRI from baseline to determine if there is a reduction of cardiac iron burden.
Time Frame: 12 months
Population: Number of participants with improvement
Measure: Count of Participants; unit: Participants
Groups:
- Deferasirox and Deferiprone Combination Chelation: Deferasirox and deferiprone
Arm/Group | Deferasirox and Deferiprone Combination Chelation
Number analyzed (Participants) | 6
Participants | 3

ADVERSE EVENTS:
Arm/Group | Deferasirox and Deferiprone
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox and Deferiprone (N=9)
viral syndrome (General disorders) | 1 (1) — Admitted with fever and abdominal pain thought unrelated to study treatment
perirectal abscess (Infections and infestations) | 1 (2) — Unrelated to study drug
Rectal bleeding from hemorrhoid (Gastrointestinal disorders) | 1 (1) — unrelated to study treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferasirox and Deferiprone (N=9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Nausea/vomiting (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
ALT elevated (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes